CLINICAL TRIAL: NCT07035925
Title: Prospective Multi-Center, Single Arm, Study Evaluating the Safety and Efficacy of an ECM Hydrogel for the Treatment of Anorectal Fistulas
Brief Title: Study Evaluating the Safety and Efficacy of an ECM Hydrogel for the Treatment of Anorectal Fistulas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECM Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECMT-100-1
Record Dates: First submitted 2025-05-13; First posted 2025-06-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Prospective Multi-Center, Single Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): ECMT-100
  Subjects will be followed for 12 months following last treatment with ECMT-100.
  Subjects are eligible for one repeat treatment as determined by the clinician/investigator at or prior to the 6-month visit.
  Interventions: Device: ECMT-100

INTERVENTIONS:
Device: ECMT-100 — Colloidal hydrogel

SUMMARY:
Safety and Efficacy of ECMT-100 for the Treatment of Anorectal Fistulas

DETAILED DESCRIPTION:
ECMT-100 is a colloidal hydrogel derived from extracellular matrix (ECM), formulated to adhere to sub-epithelial soft tissue and allow for filling of anorectal fistulas to reinforce and promote fistula tract closure. ECMT-100 is a medical device and should be administered via catheter within the fistula tract following curettage of the tract, with draining setons used preoperatively.

ECMT-100 is a mucoadhesive hydrogel composed of ECM formulated to adhere to the gastrointestinal mucosa, fill the transsphincteric fistula tract, and promote tract closure by allowing for timely host tissue integration without fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age.
* Provide informed consent
* Non-pregnant females
* Clinical diagnosis of 1 high transsphincteric anorectal fistula, with 1 internal opening and 1-2 external openings, with a single seton in place.
* Seton placement for a minimum of 3 months
* Willingness to participate in post-operative follow-up evaluations.

Exclusion Criteria:

* Inability to provide informed consent.
* Medical history of Crohn's disease/Ulcerative Colitis.
* Subjects with multiple fistula tracts (defined as >1 internal opening and/or >2 external openings), secondary tracts, horseshoe fistulas, J-pouch fistulas, superficial fistulas, ano/recto-vaginal fistulas or rectourethral fistulas.
* Previous fistulotomy/fistulectomy at the target treatment site (a history of these procedures at other locations is not exclusionary).
* Fistula of traumatic origin including obstetric.
* Evidence of ongoing local infection.
* Evidence of active abscess at the time of treatment.
* Chronic disease such as congestive heart failure, liver disease, renal disease, insulin dependent diabetes (as determined by A1C reading from past 6-12 months), or any chronic illness that may interfere with participation in this study.
* Active and unstable disease state or infection anywhere in the body per investigator's evaluation and determination.
* Autoimmune disease that is not stable.
* Subjects who are immunocompromised such as known human immunodeficiency virus (HIV) or currently receiving chemotherapy or radiation therapy.
* Ongoing use of antiplatelet drugs. Subjects may be included in the study if antiplatelet drugs have been stopped for 5 to 7 days prior to surgery.
* Known coagulopathy (demonstrated by stated or medical record history of diagnosis)
* Pregnancy
* Previous history of radiation therapy in the area of the fistula.
* History of collagen disease.
* Known allergy to porcine products.
* Religious objection to use of porcine products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2028-04-24 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months from treatment
  Number of Adverse Events

SECONDARY OUTCOMES:
Percentage of Subjects in whom external openings of the fistula have closed | 12 months from treatment
  Physical exam to confirm closure and absence of discharge
Changes in Fecal Incontinence | 12 months from treatment
  Wexner Score - Cleveland Clinic Fecal Incontinence Score; changes from baseline
Changes in Quality of Life | 12 months from treatment
  Medical Outcomes Study Questionnaire Short Form 36; changes from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania